CLINICAL TRIAL: NCT05530018
Title: Developing and Feasibility Testing of a Brief Contact Intervention to Reduce Self-harm Repetition Through Co-design.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202206137RINA
Record Dates: First submitted 2022-08-31; First posted 2022-09-07 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Suicide and Self-harm
Keywords: self-harm; psychological intervention
MeSH Terms: conditions — Suicide; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCI group (Experimental): Participants will be asked to participate in a brief contact intervention and to evaluate its feasibility, including the feasibility of recruitment, intervention resources, the appropriateness of data collection, and the acceptance of the intervention.
  Interventions: Behavioral: Brief contact intervention

INTERVENTIONS:
Behavioral: Brief contact intervention — The brief contact intervention (BCI) will send out text messages to the participants. The text messages will include caring messages, reminders of appointments, and a link to a web page. The web page is anticipated to include safety planning, volitional helpsheet, and resources information. The text messages are anticipated to send out to the participants on a weekly base for 6 weeks in a row, and then change to monthly reminders. The monthly reminders are anticipated to include caring messages, reminders of appointments, and invitations to encourage the participants to click the previous web links again. The monthly reminders are anticipated to send out to the participants three times in a row. In the final reminder, the participants will be told that this intervention is going to end. In total, the participants will receive 9 texts within 5 months.

SUMMARY:
Suicide is a major public health issue. Repeated self-harm may lead to potential future suicide deaths. In addition, it may lead to substantial loss in medical costs. Recently, smartphones have been widely used. Researchers started to apply mobile health to support individuals with self-harm experiences and to combine brief contact interventions which require lower cost to reduce repeated self-harm. However, the research evidence remains sparse. Furthermore, self-harm behaviors might be influenced by different cultural contexts. There is a need to conduct local studies in Taiwan. The aim of this study is to establish a co-design team which includes service users and service providers, to collaboratively develop a text- and web-based brief contact intervention (BCI) to reduce repeated self-harm, and to evaluate the feasibility of the intervention.

DETAILED DESCRIPTION:
Study objectives:

1. To establish a co-design team and develop a brief contact intervention (BCI), including the content, frequency, settings, and outcome measures of the intervention.
2. To evaluate the feasibility of BCI, including the feasibility of recruitment, required resources, the appropriateness of data collection, and the acceptability of the BCI.

Methods:

1. In study 1, we will recruit 4-6 service users and 4-6 service providers respectively, and we will conduct focus groups to discuss the content of the BCI. We will conduct individual interviews with participants to explore their experiences and perspectives regarding their participation in the co-design team.
2. In study 2, we will recruit 30 participants who have self-harm experiences to participate in the BCI. The BCI will be delivered through texts and web pages and will last around 5 months. The content of BCI will include caring messages, reminders of appointments, safety planning, volitional help sheet, and resources information. We will collect user engagement data and compare study outcomes (e.g., suicidal ideation and behaviors, brief symptom rating scale (BSRS), and mental well-being scale) before and after receiving the BCI. We will collect the participants' feedback regarding the BCI and evaluate the required resources to further revise the BCI.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years or over
* Mentally and physically stable and able to participate in individual interviews and interventions
* Able to communicate in Mandarin and provide written informed consent
* Willing to be recorded during the interviews
* Received medical treatments or aftercare due to self-harm experiences, including self-harm ideations, self-harm behaviors, suicidal ideations, and suicidal attempts.
* Able to use the smartphone to access the internet

Exclusion Criteria:

* Mental and physical states are unstable (e.g., unconscious, severe psychiatric symptoms, strong suicidal ideations with specific suicide plans) to complete the interviews and interventions according to the health professionals.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
The acceptability of the intervention to participants | within 3 months of study completion
  The investigators will conduct face-to-face qualitative interviews to understand the acceptability of the intervention amongst participants.
The feasibility of intervention to participants | within 3 months of study completion
  The investigators will conduct face-to-face qualitative interviews to understand the feasibility of intervention amongst participants.
Participant recruitment | through study completion, an average of 1 year
  Recruitment: the proportion of participants who are eligible and invited actually consent to participate.
Participant retention rate | 3 month
  The proportion of participants who can be reached by in-person or phone contact at the 3 month follow-up.
Participant retention rate | 6 month
  The proportion of participants who can be reached by in-person or phone contact at the 6 month follow-up.
Number of repeated self-harm episodes (self-report) | 3 month
  Number of repeated self-harm episodes per person at 3 month after intervention based on self-report.
Number of repeated self-harm episodes (self-report) | 6 month
  Number of repeated self-harm episodes per person at 6 month after intervention based on self-report.
Number of repeated self-harm episodes (nationwide self-harm registry) | 3 month
  Number of repeat self-harm episodes per person at 3 month after intervention recorded in the nationwide self-harm registry
Number of repeated self-harm episodes (nationwide self-harm registry) | 6 month
  Number of repeat self-harm episodes per person at 6 month after intervention recorded in the nationwide self-harm registry

SECONDARY OUTCOMES:
Self-Efficacy to Avoid Suicidal Action (SEASA) | From enrollment to 3 months and 6 months
  Access participants' self-efficacy and stages of change in relation to suicide ideation and attempt at baseline/3/6 month.
  The total score ranges from 0 to 24, with a score of 24 indicating the highest self-efficacy in controlling suicidal thoughts.
Help-seeking behavior questionnaire | From enrollment to 3 months and 6 months
  Assess the help-seeking behaviours of participants at baseline/3/6 month. The total score ranges from 0 to 9, with a score of 9 indicating the highest level of help-seeking behaviors (knowing how to help oneself and where to access resources).
Brief Symptom Rating Scale (BSRS) | From enrollment to 3 months and 6 months
  Briefly evaluate the psychological distresses of participants at baseline/3/6 month.
  The total score ranges from 0 to 25. Categorized as "mild" with score 6-9, "moderate" with score 10-14, and "severe" with score more than 15.
The World Health Organisation- Five Well-Being Index (WHO-5) | From enrollment to 3 months and 6 months
  Measure the current mental wellbeing of participants at baseline/3/6 month. The total score ranges from 0 to 25, with a score of 25 indicating the best quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Sen Chang, MD, MSc, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan